CLINICAL TRIAL: NCT04447703
Title: Technology-Enhanced Acceleration of Germline Evaluation for Therapy - The TARGET Study
Brief Title: Technology-Enhanced Acceleration of Germline Evaluation for Therapy, TARGET Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20G.013; 19CHAL05 (Other Grant/Funding Number: Prostate Cancer Foundation); JT 14902 (Other: JeffTrial Number)
Record Dates: First submitted 2020-04-23; First posted 2020-06-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interviews as Topic; Genetic Counseling; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aim I (Interview) (Experimental): Providers attend an interview over 1 hour to discuss how they would use the tool, then receive the tool to test in their clinic for 2 weeks. After 2 weeks, providers discuss their experience using the tool over 10-15 minutes. Providers have the option to use the tool for up to 6 months and complete a brief survey about the benefits and limitations of the tool for patient identification in Arm II.
  Interventions: Other: Interview; Other: Internet Based Intervention; Other: Survey Administration
- Aim II: Arm I (Genetic Counseling, Genetic Testing) (Active Comparator): Patients receive genetic counseling with a certified genetic counselor in-person, by telehealth, or over the phone (according to patient preference). Patients may then undergo genetic testing.
  Interventions: Other: Genetic Counseling; Genetic: Genetic Testing; Other: Survey Administration
- Aim II: Arm II (WBGE, Genetic Couseling, Genetic Testing) (Experimental): Patients receive a link to the web-based genetic education tool online including all elements of genetic counseling in written modules and in a series of professional videos. Patient may then undergo genetic testing. Patient may cross-over to Arm I to see a genetic counselor.
  Interventions: Other: Genetic Counseling; Other: Internet-Based Intervention; Genetic: Genetic Testing; Other: Survey Administration

INTERVENTIONS:
Other: Interview — Attend Interview
  Arms: Aim I (Interview)
Other: Internet Based Intervention — Use web-based genetic education tool online
  Arms: Aim I (Interview)
Other: Survey Administration — Ancillary Studies
  Arms: Aim I (Interview)
Other: Genetic Counseling — Receive in-person, telehealth, or over-the-phone genetic counseling
  Arms: Aim II: Arm I (Genetic Counseling, Genetic Testing)
Genetic: Genetic Testing — Undergo genetic testing
  Other Names: Genetic Analysis, Genetic Examination, Genetic Test, Genetic Testing, Genetic Testing
  Arms: Aim II: Arm I (Genetic Counseling, Genetic Testing)
Other: Survey Administration — Ancillary Studies
  Arms: Aim II: Arm I (Genetic Counseling, Genetic Testing)
Other: Genetic Counseling — Receive in-person, telehealth, or over-the-phone genetic counseling
  Arms: Aim II: Arm II (WBGE, Genetic Couseling, Genetic Testing)
Other: Internet-Based Intervention — Use web-based genetic education tool online
  Arms: Aim II: Arm II (WBGE, Genetic Couseling, Genetic Testing)
Genetic: Genetic Testing — Undergo genetic testing
  Other Names: Genetic Analysis, Genetic Examination, Genetic Test, Genetic Testing, Genetic Testing
  Arms: Aim II: Arm II (WBGE, Genetic Couseling, Genetic Testing)
Other: Survey Administration — Ancillary Studies
  Arms: Aim II: Arm II (WBGE, Genetic Couseling, Genetic Testing)

SUMMARY:
This trial performs user testing of a mobile-friendly patient history collection and genetic education tool to improve healthcare providers' understanding of prostate cancer genetic testing. This trial also compares traditional genetic counseling versus a web-based genetic education (WBGE) tool to provide information about genetic testing to men with prostate cancer. The WBGE tool has educational modules on genetic counseling and testing, as well as a patient history collection tool to help providers learn which patients may carry genetic mutations and may be considered for genetic counseling and genetic testing. The purpose of this research is to use technology to deliver information on genetic testing for prostate cancer to patients to help them decide whether or not to receive genetic testing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Perform user-testing of an education and patient history collection mobile tool among medical oncologists, radiation oncologists, and urologists across study practice settings, including Veterans Affairs to address genetic referral needs (n=10 providers). (Provider-focused) II. Develop multimedia web-based pretest genetic education (WBGE) tool and conduct a randomized trial of traditional genetic counseling (GC) (Arm 1) versus (vs.) WBGE (Arm 2) for informed and timely uptake of genetic testing for men with lethal/predicted lethal prostate cancer (PCA). (Patient-focused)

OUTLINE:

AIM I: Providers attend an interview over 1 hour to discuss how they would use the tool, then receive the tool to test in their clinic for 2 weeks. After 2 weeks, providers discuss their experience using the tool over 10-15 minutes. Providers have the option to use the tool for up to 6 months and complete a brief survey about the benefits and limitations of the tool for patient identification in Arm II.

AIM II: Patients are randomized to 1 of 2 arms.

ARM I (TRADITIONAL GENETIC COUNSELING): Patients receive genetic counseling with a certified genetic counselor in-person, by telehealth, or over the phone (according to patient preference). Patients may then undergo genetic testing.

ARM II (WEB-BASED GENETIC EDUCATION): Patients receive a link to the web-based genetic education tool online including all elements of genetic counseling in written modules and in a series of professional videos. Patients may then undergo genetic testing. Patients may cross-over to Arm I to see a genetic counselor.

After the completion of study, patients are followed up yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria

* AIM 1: Medical oncologists, radiation oncologists and urologists spanning Veterans Affairs (VA), academic, and community settings
* AIM 2: Any English speaking man >= 18 with PCA who has computer and web-access and meets any one of the following:

  * Metastatic disease
  * T3a or higher
  * Prostate specific antigen (PSA) > 20
  * Grade group 4 or higher
  * Intraductal or cribriform histology
  * Biochemical recurrence
  * Ashkenazi Jewish ancestry
  * Family history criteria (see below) ** Family history: If any one of the following levels are met, the person is eligible:

    * Level 1: >= 1 close blood relative (first degree relative [FDR], second degree relative [SDR], third degree relative [TDR]) diagnosed with breast cancer =< age 50 or the following cancers at any age: pancreatic, ovarian, or metastatic or intraductal/cribriform prostate cancer
    * Level 2: >= 2 close blood relatives (FDR, SDR, TDR) on same side of the family with breast or prostate cancer at any age
    * Level 3: one brother, father, or >= 2 family members (close blood relatives - FDR, SDR, TDR) on the same side of the family diagnosed with prostate cancer at < 60
    * Level 4: >= 3 cancers on the same side of the family (especially if diagnosed =< 50): bile duct, breast, colorectal, endometrial, gastric, kidney, melanoma, ovarian, pancreatic, prostate (grade groups 2-5 if known), small bowel, or urothelial

Exclusion Criteria

* Age < 18 years
* Mental or cognitive impairment that interferes with ability to provide informed consent
* Non-English speaking
* Having had prior germline genetic testing for inherited cancer risk (pertains to aim 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
User Testing of the Provider Tool - (Aim I) | Up to 6 months
  Provider perspectives will include: (1) whether the target population can use the tool in the way it was intended (i.e., to perform patient history collection to determine consideration for germline testing), and (2) interaction with this tool affects the user's cognitive representation of genetic testing for prostate cancer (PCA). To evaluate the first point, will collect initial information from participants regarding their experience with the guidelines for genetic testing and how they collect data on family history. Will evaluate participants' mental model for germline testing and how they identify suitable candidates before interaction with the tool. Will use a cognitive concept mapping technique, which can be used to formalize a person's cognitive representation for complex topics. Feedback from this testing will be used to iteratively refine the tool while it is being used by providers to identify patients randomized trial in Aim II.
Decisional Conflict (Aim II) | Up to 6 months
  Will be assessed for non-inferiority between study arms. Evaluated using the O'Connor decisional conflict scale, which captures sub-scores over 16-questions for uncertainty, feeling of being informed, values clarity, support, and effective decision making on a 5-point Likert scale

SECONDARY OUTCOMES:
Cancer Genetics Knowledge (Aim II) | Up to 6 Months
  Assessed using pre- and post-intervention surveys. Cancer genetics knowledge will be adapted from Erblich. et al (2005) for relevance to PCA genetics (23 True/False questions) (Cronbach's alpha = 0.92).
Genetic Testing Uptake (Aim II) | Up to 5 years
  Assessed using pre-and post-intervention surveys
Satisfaction with Genetic Counseling or Web-Based Genetic Education (Aim II) | After viewing the web tool
  Will capture men's satisfaction with each arm using the Satisfaction with Genetic Counseling Scale at the end of pre-test genetic counseling or after viewing the web tool. This 6-item scale includes questions such as: "My genetic counselor seemed to understand the stresses I was facing," and "The genetic counseling session was valuable to me" rated on a 5-point Likert scale (Cronbach's alpha 0.7-0.88). The questions will be adapted for web-based pretest genetic education such as "This webtool addressed all of the concerns I had" or "The webtool was valuable to me".

OTHER OUTCOMES:
Understanding of personal genetic test results (Aim II) | Up to 5 years
  Assessed using pre- and post-intervention surveys.
Sharing of genetic information with families (Aim II) | Up to 5 years
  Assessed using pre- and post-intervention surveys.
Literacy (Aim II) | Up to 5 years
  Assessed using pre- and post-intervention surveys.
Numeracy (Aim II) | Up to 5 years
  Assessed using pre- and post-intervention surveys.
Diet (Aim II) | Up to 5 years
  Assessed using pre- and post-intervention surveys.
Physical activity (Aim II) | Up to 5 years
  Assessed using pre- and post-intervention surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Veda Giri, MD, Principal Investigator — Clinical Cancer Genetics Yale School of Medicine; Stacy Loeb, MD, MSc, Principal Investigator — NYU- Langone Health, Manhattan VA Hospital
Locations (5):
- United States (5):
  - VA New York Harbor Health System- Manhattan Campus, New York, New York
  - New York University- Langone Health, New York, New York
  - Associated Medical Professions of New York, Syracuse, New York
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Washington/ SCCA, Seattle, Washington

REFERENCES:
- [Derived] Loeb S, Keith SW, Cheng HH, Leader AE, Gross L, Sanchez Nolasco T, Byrne N, Hartman R, Brown LH, Pieczonka CM, Gomella LG, Kelly WK, Lallas CD, Handley N, Mille PJ, Mark JR, Brown GA, Chopra S, McClellan A, Wise DR, Hollifield L, Giri VN. TARGET: A Randomized, Noninferiority Trial of a Pretest, Patient-Driven Genetic Education Webtool Versus Genetic Counseling for Prostate Cancer Germline Testing. JCO Precis Oncol. 2024 Mar;8:e2300552. doi: 10.1200/PO.23.00552. PMID 38452310
- [Derived] Loeb S, Cheng HH, Leader A, Gross L, Nolasco TS, Byrne N, Wise DR, Hollifield L, Brown LH, Slater E, Pieczonka C, Gomella LG, Kelly WK, Trabulsi EJ, Handley N, Lallas CD, Chandrasekar T, Mille P, Mann M, Mark JR, Brown G, Chopra S, Wasserman J, Phillips J, Somers P, Giri VN. Technology-enhanced AcceleRation of Germline Evaluation for Therapy (TARGET): A randomized controlled trial of a pretest patient-driven webtool vs. genetic counseling for prostate cancer germline testing. Contemp Clin Trials. 2022 Aug;119:106821. doi: 10.1016/j.cct.2022.106821. Epub 2022 Jun 14. PMID 35710085